CLINICAL TRIAL: NCT00994513
Title: Effect of Alpha Lipoic Acid on Obesity Related Comorbidities
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Xinjiang Medical University (Other)
Responsible Party: Xiaoling Wang, Assistant Professor, Medical College of Georgia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HAC08-07-02
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Obesity; Cardiovascular Disease; Type 2 Diabetes
Keywords: Antioxidant; Obesity
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Diabetes Mellitus, Type 2 | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALA (Active Comparator): alpha lipoic acid 1200 mg/day
  Interventions: Dietary Supplement: Alpha Lipoic Acid
- Placebo (Placebo Comparator): placebo 1200 mg/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Alpha Lipoic Acid — 1200 mg/day
  Other Names: Lipoic acid
  Arms: ALA
Dietary Supplement: Placebo — 1200 mg/day
  Arms: Placebo

SUMMARY:
The major objective of this study is to conduct a double-blind, placebo-controlled, randomized clinical trial to assess whether oral alpha lipoic acid supplementation will decrease cardiovascular disease and type 2 diabetes risk in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Han ethnicity
* BMI≥25kg/m2
* Having at least one of the following risk factors: borderline hypertension (130mmHg≤SBP<140mmHg or 85mmHg≤DBP<90mmHg), dyslipidemia (fasting total cholesterol ≥240mg/dl or HDL-C<40mg/dl), or impaired fasting glucose (fasting glucose levels between 6.1 and 7.0mmol/L)
* 18-60 years old
* Not on any antioxidant vitamin supplement

Exclusion Criteria:

* Pregnancy, lactation or child-bearing age without birth control device
* History of hypertension, diabetes, coronary heart disease(CHD), cancer or liver disease
* Anything that would impede the subject from complying with the ALA treatment
* History of psychiatric problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Biomarkers of oxidative stress | 2 months
Insulin sensitivity | 2 months
Endothelial function | 2 months

SECONDARY OUTCOMES:
Inflammatory markers | 2 months
Blood pressure | 2 months
Fasting lipid profile | 2 months
Pulse wave velocity | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Xinjiang Medical University, Ürümqi, Xinjiang, China